CLINICAL TRIAL: NCT06829758
Title: Effectiveness of a Community Intervention in Reducing the Feeling of Unwanted Loneliness, Social Risk, and Social Isolation in the Population Over 65 Years Old in La Palma, Focusing on Healthy Habits, Sleep Hygiene, and Digital Literacy
Brief Title: Compartiendo Salud: Community-Based Intervention for Loneliness
Acronym: SoledadLP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Collaborators: University of La Laguna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CHUC_2023_94
Record Dates: First submitted 2025-02-10; First posted 2025-02-17 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Loneliness
Keywords: Social Support; Community Health Nursing; Health Education; Aged
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): The intervention proposed (Compartiendo Salud) is a multicomponent intervention based on prevention and on promoting the health of older adults that live alone. Quasi-experimental study was designed with pre- and post- intervention (at three months) measurements, with no Control Group or randomisation.
  Interventions: Behavioral: Compartiendo Salud

INTERVENTIONS:
Behavioral: Compartiendo Salud — The intervention proposed (Compartiendo Salud) is a multicomponent intervention based on prevention and on promoting the health of older adults that live alone. The community-based intervention consists in five workshops that are carried out during a week (one day for each workshop). The sessions (which last 2.5 hours each) are designed in an expository and participatory way, using gaming dynamics that foster learning and social interaction. The content of the workshops is the same for all BHDs. Each workshop addresses risk factors that predispose the population to experiencing more unwanted loneliness and social isolation. The concepts corresponding to each of the five sessions that comprise the intervention are: Sleep hygiene, Healthy and sustainable eating habits, Physical activity and exercise, Memory and music therapy, Digital literacy

SUMMARY:
Unwanted loneliness is the gap between the social relations a person has and those they want. The main objective of this research is to assess the impact of a multidimensional community-based intervention on the feeling of unwanted loneliness in the population over the age of 65 years old, who living alone, under social risk or socially isolated living in the La Palma island.

DETAILED DESCRIPTION:
Loneliness is strongly associated with a significant impact on physical health, depression and may in fact be an independent risk factor for depression. Fur-thermore, it is negatively associated with healt problems, like higher blood pressure, poorer sleep, immune responses to stress, and poorer cognition over time in the elderly. The absence of personal connections is related to the adoption of worse life habits and to increased morbidity, with the consequent higher risk of suf-fering cardiovascular and endocrine diseases, mental health pathologies and risk of falls.

The secondary objectives proposed are as follows: Increasing the number of opportunities for social interaction during the intervention; Contributing tools to improve the participants' social skills in the intervention; Fostering self-care and healthy habits in the participants; Reducing maladaptive thoughts; Educating on sleep hygiene measures and non-pharmacological treatments.

The null hypothesis (H0) of this research is that in the population under study, the proposed multidimensional community intervention will not significantly impact the feeling of unwanted loneliness and the health management of these subjects.

ELIGIBILITY:
Inclusion Criteria:

* People over the age of 65 and living alone
* Nursing diagnosis of social risk
* Nursing diagnosis of social isolation

Exclusion Criteria:

* presenting moderate/severe cognitive decline or Pfeiffer scores above 6
* individuals with uncorrected hearing deficits that hinder group interaction
* participants not subjected to the pre- and post-interventions measurements
* participants that do not take part in at least four of the five sessions scheduled

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Feeling of unwanted loneliness | Pre- and post- intervention (at three months)
  It was measured using the "UCLA (University of California at Los Angeles) Loneliness scale" test validated in Spain. This instrument is based on three dimensions: Relational connection; Social connection; and Self-perceived isolation. It uses a 4-point scale ranging from "Never" to "Frequently" for responses 10 items. Scores above 30 correspond to "No loneliness", between 20 and 30 mean "Moderate loneliness" and less than 20 points is "Severe loneliness"

SECONDARY OUTCOMES:
Number of Participants with Social risk | Pre- and post- intervention (at three months)
  It was measured using the Gijón Social risk detection questionnaire. It assesses family and economic situations, housing, social relations and support from social networks. It uses a 5-point scale ranging from best to worse situation, for responses 5 items. Scores: Good/Acceptable social situation: from 5 to 9 points; Social risk: from 10 to 14; and social problem: more than 15
Number of Participants with Low Perceived social support | Pre- and post- intervention (at three months)
  It was measured with Duke's questionnaire. It assesses perceived social support and consists of 11 items, each one assessed with a Likert scale from 1 to 5. Scores equal to or higher than 32 indicate "Normal support", whereas less than 32 points means "Low perceived social support"
Number of Participants with Anxiety or depression | Pre- and post- intervention (at three months)
  They were assessed using Goldberg's questionnaire with two subscales: Anxiety and Depression. Each of them is structured with 4 initial screening items to determine the probability of a mental disorder and a second group with 5 items that are only formulated if positive answers are given to the screening questions (at least 2 in the Anxiety subscale and at least 1 in the Depression subscale). The type of response of the questionnaire is dichotomous (Yes/No). The cut-off points are as follows: scores equal to or higher than 4 for the Anxiety subscale; and values equal to or higher than 2 for Depression. In the geriatric population, it has been proposed to use it as a single scale, with a cut-off point equal to or higher than 6
Number of Participants with Risk of loneliness | Pre- and post- intervention (at three months)
  Nursing diagnosis "Risk of loneliness" (Yes/No) and presence/absence of each of its defining characteristics: Affective deprivation; Emotional Deprivation; Physical isolation; Social isolation.
Number of Participants with Social Isolation | Pre- and post- intervention (at three months)
  Nursing diagnosis "Social Isolation" (Yes/No) and presence/absence of each of its defining characteristics: Low social activity levels; Change in physical aspect; Explicit dissatisfaction with social connections; Social reclusion; Social behaviour inconsistent with cultural norms; Reporting feeling insecure in public; Reduced eye contact.
Number of Participants with Smoking | Pre- and post- intervention (at three months)
  The smoking assessment included in the habits module of the electronic clinical history of Primary Health Care of the Canary Islands Health Service Drago-AP will be used: Non-smoker/Smoker in undetermined phase/Smoker in pre-contemplation phase (consonant)/Smoker in contemplation phase (dissonant)/Smoker in preparation phase/Smoker in action phase/Smoker in maintenance phase/Former smoker since 1-10 years/Former smoker since more than 10 years/Passive smoker
Number of Participants with alcoholism | Pre- and post- intervention (at three months)
  The alcoholism assessment included in the habits module of the electronic clinical history of Primary Health Care of the Canary Islands Health Service Drago-AP will be used: Non-drinker/Moderate drinker/Risk drinker/Drinking problem
Number of Participants without sleep problems | Pre- and post- intervention (at three months)
  Sleep problem (Yes/No)
Number of Participants with caregiver | Pre- and post- intervention (at three months)
  Dichotomous variables (Yes/No)
Number of Participants belonging to an organized group | Pre- and post- intervention (at three months)
  Dichotomous variables (Yes/No)
Number of Participants what does it feel like Integrated in the area where they live | Pre- and post- intervention (at three months)
  Dichotomous variables (Yes/No)
Number of Participants with Activities in free and/or leisure time | Pre- and post- intervention (at three months)
  Dichotomous variables (Yes/No)
Number of Participants with Home-based care; Social assistance | Pre- and post- intervention (at three months)
  Dichotomous variables (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Alba Francisco-Sánchez, Nursing Specialist, Principal Investigator — Atención Primaria. Área de Salud de La Palma. Servicio Canario de Salud
Locations (1):
- La Palma Health Area. Canary Islands Health Service., Santa Cruz de La Palma, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon reasonable request. The data to be shared will include all IPD that underlie results in a publication, as well as the statistical analysis plan, informed consent form and the analytic code.
  All sensitive data will be anonymized to ensure the privacy and confidentiality of the participants.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The complete IPD will be available for sharing six months after the study's conclusion.
Access Criteria: As an access criterion for Individual Participant Data (IPD), it is required that no information be requested that could compromise the anonymity of participants. This ensures adherence to ethical research standards and the protection of personal data, safeguarding the confidentiality and privacy of all individuals involved.